CLINICAL TRIAL: NCT07151950
Title: Obi Medical Robot: Evaluating Effectiveness Related to Usability in Providers, Caregivers & Patients
Brief Title: Obi Medical Robot: Evaluating Effectiveness Related to Usability
Status: Active, not recruiting | Type: Observational
Sponsor: Desin LLC (Industry)
Collaborators: The Driving Doctor: Adaptive Driving & Rehabilitation Solutions, PC (Other)
Responsible Party: Principal Investigator, Andrea Fairman, Principal Investigator & Research Consultant, The Driving Doctor: Adaptive Driving & Rehabilitation Solutions, PC
Other Study IDs: IFD-DES-081
Record Dates: First submitted 2025-08-12; First posted 2025-09-03 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Upper Extremity Impairments; Cerebral Palsy (CP); ALS - Amyotrophic Lateral Sclerosis; Rett Syndrome
Keywords: upper extremity impairments; Robot Assisted Feeding; assistive technology; usability
MeSH Terms: conditions — Cerebral Palsy; Amyotrophic Lateral Sclerosis; Rett Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (3):
- Providers who recommend Obi
- Caregivers of Persons who trial Obi: Caregivers who assist persons with disabilities who trial Obi are invited to share their perspectives and experiences in helping to set up the device, interpret instructions, and describe the experience of trialing Obi from their perspective as a caregiver
  Interventions: Device: One-week trial of Obi Medical device, which provides robotic assistance with feeding to persons with upper extremity impairments who are unable to self-feed in the traditional manner using utensils
- Persons with Disabilities who trial Obi
  Interventions: Device: One-week trial of Obi Medical device, which provides robotic assistance with feeding to persons with upper extremity impairments who are unable to self-feed in the traditional manner using utensils

INTERVENTIONS:
Device: One-week trial of Obi Medical device, which provides robotic assistance with feeding to persons with upper extremity impairments who are unable to self-feed in the traditional manner using utensils — This study explores the stakeholders' experiences in recommending and using Obi. Stakeholders/Participants include:
  1. Persons with disabilities or conditions which prevent them from successfully using their upper extremities (UE) to self-feed independently
  2. Caregivers of the persons with disabilities described above
  3. Providers (OT, SLP, PT, ATP, etc.) who provide services to persons with disabilities
  Groups: Caregivers of Persons who trial Obi; Persons with Disabilities who trial Obi

SUMMARY:
This mixed-methods usability study evaluates the effectiveness of the Obi Gen 3 robotic feeding device in meeting user needs among providers, caregivers, and patients. Participants will complete a one-week trial using Obi in home, school, or community settings, followed by feedback surveys and optional interviews. The study seeks to validate that the device design meets usability requirements prior to broader deployment.

DETAILED DESCRIPTION:
The study assesses the usability of Obi Gen 3 through quantitative surveys and qualitative interviews across three user groups: providers, caregivers, and patients. Measures include the System Usability Scale (SUS), questions based on the Matching Person & Technology (MPT) assessment and framework, and a custom Obi Medical Device Needs Assessment (MDNA). Data collection includes pre-trial in-office screening and post-trial surveys gathered remotely using Qualtrics. Optional follow-up interviews gather further feedback. The study aims to verify that the Obi Gen 3 meets its intended use and user needs in real-world environments.

ELIGIBILITY:
Inclusion Criteria:

* Providers with relevant expertise to recommend and evaluate patients' ability to use Obi
* Caregivers directly assisting users with Obi
* Adults or children (≥5 years) needing assistive feeding technology to self-feed

Exclusion Criteria:

* Inability to provide informed consent/assent
* Cognitive impairments that may prevent the ability to understand or respond to the survey questions
* Non-English speakers (English-only materials)
* Residents of California who are new Obi users

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study will enroll three key stakeholder groups to evaluate the usability of the Obi Gen 3 device:
  Pediatric and Adult Patients - Individuals aged 5 years and older with functional self-feeding impairments who are recommended for Obi use by a clinician. Patients must have sufficient cognitive and communication abilities to provide feedback directly or with assistance.
  Caregivers - Family members or paid support personnel who assist the patient with meals or device operation. Caregivers will provide insight into the impact of the device on mealtime routines, supervision needs, and caregiving burden.
  Clinicians/Providers - Healthcare professionals (e.g., occupational therapists, speech-language pathologists, rehabilitation specialists) who assess, recommend, or train patients in Obi use. Providers will evaluate device usability, safety, and integration into clinical practice.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2025-05-10 (Actual); Primary Completion 2025-08-12 (Actual); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
System Usability Scale | one week post trial
  The System Usability Scale (SUS) is a widely used, reliable tool for measuring the usability of a product or system. It consists of a 10-item questionnaire with a five-point Likert scale ranging from "Strongly Disagree" to "Strongly Agree." SUS provides a single score on a scale from 0 to 100 that reflects the overall ease of use and user satisfaction. Developed by John Brooke in 1986, the SUS is technology-agnostic and can be applied across a wide range of systems, including software, websites, and assistive technologies. Its simplicity, robustness, and versatility make it a standard in usability evaluation.
Non-Standardized, Custom Survey | one week trial
  Another primary outcome for this study is stakeholder-reported usability of the Obi Gen 3 device, as assessed by structured, study-specific surveys developed for this clinical investigation. Separate but parallel survey instruments were created for patients, caregivers, and clinicians/providers to capture device performance and user experience from multiple perspectives. Each survey includes both closed-ended and open-ended questions addressing:
  * Ease of use - learning to operate the device, understanding controls, and integrating it into mealtime routines
  * Effectiveness - ability to self-feed, control bite timing and size, and accommodate a variety of foods
  * Satisfaction - overall impressions, perceived benefits, and willingness to recommend the device
  * Safety and comfort - perceived safety during operation, confidence in device reliability, and comfort while using the device
  * Suggestions for improvement - opportunities for design or functionality enhancements
Functional Eating Status | One week trial
  Functional eating status is measured by the clinical provider at baseline (without use of Obi) and again one week post-trial (with use of Obi). The participants' level of performance is assessed on a Likert Scale as follows: 0 - No problem, 1 - Mild, 2 - Moderate, 3 - Severe, 4 - Complete

CONTACTS AND LOCATIONS:
Locations (1):
- Desin, Llc, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared due to the small sample size, the vulnerability of the pediatric population, and the inclusion of potentially identifiable health information. Data will be reported only in aggregate form to protect participant privacy and comply with applicable privacy regulations (e.g., HIPAA).

DOCUMENTS (2):
  • Study Protocol (2025-04-11): https://cdn.clinicaltrials.gov/large-docs/50/NCT07151950/Prot_000.pdf
  • Informed Consent Form (2025-04-23): https://cdn.clinicaltrials.gov/large-docs/50/NCT07151950/ICF_001.pdf